CLINICAL TRIAL: NCT07247136
Title: Study of 30-Minute Stimulation With the Neuspera Sacral Neuromodulation (SNM) System in Patients With Symptoms of Urinary Urgency Incontinence (UUI)
Brief Title: Study of 30-Minute Stimulation With the Neuspera Sacral Neuromodulation (SNM) System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neuspera Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Neuspera Medical (NSM-006)
Record Dates: First submitted 2025-11-19; First posted 2025-11-25 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Urinary Urge Incontinence
MeSH Terms: conditions — Urinary Incontinence, Urge

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Neuspera Implantable Sacral Nerve Stimulation System (Other): Implantation of the stimulator to assess effectiveness with shorter duration of stimulation
  Interventions: Device: Neuspera Implantable Sacral Neuromodulation System

INTERVENTIONS:
Device: Neuspera Implantable Sacral Neuromodulation System — Stimulation of the Sacral Nerve

SUMMARY:
Single-arm study conducted in participants for the treatment of urinary urge incontinence in patients who have failed, could not tolerate, or were not a candidate for more conservative treatments.

The objective of the study is to assess the effectiveness of 30-minutes daily therapeutic stimulation with the Neuspera System.

DETAILED DESCRIPTION:
The study is intended to investigate the potential for controlling UUI symptoms with thirty minutes of stimulation per day.

Subjects will be enrolled in a single-arm study and followed for 6 months post implant. Subjects will undergo a trial stimulation period, followed by a permanent implant. If subjects do not receive appropriate benefits with the shorter duration of stimulation, they can increase the duration of stimulation anytime as needed. Subjects may also decrease stimulation after one month to 15 minutes per day if desired.

Up to 20 subjects will be implanted.

ELIGIBILITY:
Inclusion Criteria:

* Is male or female 22 years of age or older.
* Has a diagnosis of UUI for greater than or equal to 6 months prior to the screening baseline visit date.
* Has failed, could not tolerate (stopped taking medication due to lack of efficacy or intolerable side effects), or not a good candidate for (as determined by treating physician) at least one (1) antimuscarinic or β3 adrenoceptor agonist medication.
* Is willing and able to washout (at least five half-lives) from OAB medications for a period determined appropriate based on type of OAB medication prior to the baseline bladder diary and remain off OAB medications through the study duration OR must be willing to maintain medication through the study duration.
* Has a diagnosis of UUI with at least 4 UUI episodes on a 72-hour diary.
* Has a positive stimulation trial with a 50% reduction in UUI episodes.

Exclusion Criteria:

* Has a contraindication for the Neuspera SNM System per the device labeling.
* Has a hemoglobin A1c of >8%.
* Has glucosuria.
* Has diabetic neuropathy.
* Has interstitial cystitis or bladder pain syndrome as defined by either American Urological Association (AUA) or European Association of Urology (EAU) guidelines, chronic pelvic pain, or recurrent symptomatic urinary tract infections.
* Has skin, orthopedic, neurological, or hematological (bleeding disorder) or anatomical limitations that could prevent successful placement of the neurostimulator.
* Has broken, blistered skin or compromised circulation in the area of the neurostimulator implant.
* Has neurogenic bladder dysfunction such as traumatic or atraumatic myelopathy, multiple sclerosis, Parkinsonism, or history of cerebrovascular accident.
* Has documented urinary retention within 6 months prior to the screening baseline visit date.
* Has clinically significant bladder outlet obstruction.
* Is currently undergoing or has previously undergone pelvic irradiation.
* Is a subject with a mechanical obstruction such as benign prostatic hypertrophy, urethral stricture, or cancer.
* Has current grade 3 or 4 pelvic organ prolapse including cystocele, rectocele, enterocele, procidentia or vaginal vault prolapse.
* Has received tibial nerve stimulation (TNS) in the past 3 months for the treatment of overactive bladder or unwilling to stay off TNS therapy for the study duration.
* Has received treatment of urinary symptoms with any botulinum neurotoxin type-A (BoNT-A) agent in the past 6 months; (e.g. obotulinumtoxinA, Botox,® abobotulinumtoxinA, Dysport® IncobotulinumtoxinA, Xeomin®).
* Is a woman who is pregnant or planning to become pregnant during this clinical study or is a woman of child-bearing potential who is not using a medically acceptable method of birth control. Women of child-bearing potential must undergo a pregnancy test, with clear negative result.
* Has previously had SNM therapy.
* Has active implantable medical devices such as neurostimulators, drug pumps, pacemakers, or internal defibrillators since compatibility has not been assessed.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint- Proportion of Subjects experiencing a device- and/or procedure-related AEs | 6 months
  Proportion of Subjects experiencing a device- and/or procedure-related Adverse events
Primary Effectiveness Endpoint-Percentage of all implanted subjects who experience an improvement in UUI episodes. | 1, 3 and 6 months post implant
  Percentage of all implanted subjects who experience an improvement in UUI episodes of at least 50% or more, relative to the number of UUI episodes at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Reub, MD, Principal Investigator — Southern Urogynecology
Locations (1):
- Southern Urogynecology, LLC, West Columbia, South Carolina, United States

REFERENCES:
- See also: Neuspera Medical web page — http://neuspera.com